CLINICAL TRIAL: NCT05565417
Title: A Phase 1/2a, First-in-Human (FIH), Open-Label, Dose-Escalation and Dose Expansion Study of the Monoclonal Antibody IMT-009 in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Study of the Monoclonal Antibody IMT-009 in Patients With Advanced Solid Tumors or Lymphomas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunitas Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMT-009-101
Record Dates: First submitted 2022-09-23; First posted 2022-10-04 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Triple Negative Breast Cancer; Cutaneous Squamous Cell Carcinoma; Hormone Receptor Positive Breast Carcinoma; Small Bowel Cancer; Esophageal Cancer; Colorectal Cancer; Diffuse Large B Cell Lymphoma; Hodgkin Lymphoma; Burkitt Lymphoma; Follicular Lymphoma
Keywords: Solid Tumor; Lymphoma; CD161; Non small cell lung cancer; Head and neck squamous cell carcinoma; Triple negative breast cancer; Cutaneous squamous cell carcinoma; Hormone receptor positive breast cancer; Small bowel carcinoma; Esophageal cancer; Colorectal cancer; Diffuse large B-cell lymphoma; Hodgkin lymphoma; Burkitt lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- IMT-009 Dose Escalation (Experimental): Participants will receive an assigned dose level of IMT-009 monotherapy in dose escalation. Up to 64 Participants will be enrolled in the Phase 1 portion of the study.
  Interventions: Drug: IMT-009
- IMT-009 Phase 1b (Experimental): Participants will receive an assigned dose level of IMT-009 in combination with standard of care fruquintinib. Approximately 18 Participants will be enrolled in the Phase 1b portion of the study.
  Interventions: Drug: IMT-009; Combination Product: Fruquintinib
- IMT-009 Phase 2a Cohort (s) (Experimental): Each Cohort will evaluate IMT-009 monotherapy in up to 25 Participants
  Interventions: Drug: IMT-009

INTERVENTIONS:
Drug: IMT-009 — Participants will receive an IV infusion of IMT-009 on Day 1 during each 21-day cycle.
Combination Product: Fruquintinib — Fruquintinib will be administered according to the FDA-approved United States Prescribing Information (USPI).
  Other Names: fruzaqla
  Arms: IMT-009 Phase 1b

SUMMARY:
This is a Phase 1/2a open-label, multicenter, dose escalation and dose expansion trial in which IMT-009 will be administered by the intravenous (IV) route to participants with solid tumors or lymphomas.

The main goals of this study are to:

* Find the recommended dose of IMT-009 that can be safely given to participants
* Learn more about the side effects of IMT-009
* Learn more about pharmacokinetics of IMT-009
* Learn more about the effectiveness of IMT-009
* Learn more about different pharmacokinetic biomarkers and how they might change in the presence of IMT-009

DETAILED DESCRIPTION:
IMT-009 is an Fc-attenuated monoclonal antibody that binds with high affinity and selectivity to CD161, a receptor that is broadly expressed on NK and a subset of memory T cells, blocking interactions between the receptor and its cognate ligand, CLEC2D, which is expressed on the surface of both cancer cells and immune cells. Preclinical data confirm that CD161 blockade with IMT-009 results in enhanced anti-tumor activity. This is a Phase 1/2a, open label dose escalation study of IMT-009, a fully human monoclonal antibody targeting CD161, given as a single agent in Phase 1 and potentially in combination with other antineoplastic agents in Phase 2.

ELIGIBILITY:
Key Inclusion Criteria:

Phase 1:

1. Males and females ≥18 years of age at the time of consent
2. Willingness and capacity to provide written consent
3. Patients who have histologically or cytologically-documented, unresectable locally advanced, or metastatic solid malignancy or designated lymphoma that is progressing or has failed the therapies listed below or who are intolerant of or are ineligible for or refuse standard of care therapy as detailed below.

   * Patients previously pre-treated with a checkpoint inhibitor must be anti-PD-L1 relapsed/refractory defined as having clear evidence of radiologic or clinical progression while on or within 4 months of their last anti-PD-L1 dose.
   * There is no limit to the number of prior treatment regimens a patient may have had prior to enrollment.

   Has one of the following solid tumor or lymphoma indications:
   * Non-small cell lung cancer (NSCLC) - squamous or non-squamous:

     * Must have received prior chemotherapy and a checkpoint inhibitor (either sequentially or in combination) per PD-L1 status
     * Must not have a documented EGFR, ALK, ROS, RET, BRAFV600E, Met exon 14 skipping, KRAS mutation
   * Head and neck squamous cell carcinoma (HNSCC) -- HPV+ or - :

     * Must have received prior treatment with a platinum-based chemotherapy and a checkpoint inhibitor (either sequentially or in combination) per PD-L1 status
   * Triple negative breast cancer (TNBC):

     * Must have received prior treatment with chemotherapy (anthracycline, and/or taxanes, and/or platinum, and/or gemcitabine); sacituzumab govitecan; a checkpoint inhibitor if PD-L1+; a PARPi for patients with gBRCA mutations
   * Cutaneous squamous cell carcinoma:

     * Must have received prior treatment with a checkpoint inhibitor
   * Hormone receptor positive (HR+) breast cancer:

     - Must have received endocrine therapy, a CDK 4/6 inhibitor (preferably in combination with endocrine therapy in the 1st line or 2nd line setting or as monotherapy), a PI3K inhibitor and endocrine therapy for tumors with PIK3CA activating mutation; and a PARPi for patients with gBRCA mutations
   * Small bowel carcinoma:

     * Must have received prior treatment with at least one 5FU or capecitabine based regimen (such as but not limited to FOLFOX, FOLFIRI or CAPOX) with or without bevacizumab, and a PD1/PD-L1 inhibitor alone or in combination with CTLA4 inhibitor (for MSI-H or dMMR tumors)
   * Esophageal cancer:

     * Must have received prior treatment with a platinum-based chemotherapy and a checkpoint inhibitor (either sequentially or in combination per PD-L1 status), and an anti-HER2 agent for patients with known HER2 overexpressing tumors
   * Colorectal cancer (MSS & MSI-H/dMMR):

     * Must have received at least one 5FU chemotherapy-based regimen, with bevacizumab or cetuximab/panitumumab, and / or a PD1/PD-L1 (single agent or combination with CTLA4) for dMMR/MSI-H tumors
     * For patients with known BRAF V600E mutation: must have received prior treatment with a combination of encorafenib and cetuximab or panitumumab
   * Histologically confirmed diffuse large B cell lymphoma (DLBCL)

     * Must have received at least 2 prior lines of therapy including prior treatment with chemotherapy and an anti-CD20 antibody (ie, CHOP)
     * Must be ineligible or refuse therapies with demonstrated clinical benefit such as for example CAR-T or autologous stem cell transplant
   * Hodgkin lymphoma:

     - Must have received at least 3 prior systemic therapies, including combination chemotherapy (ie, ABVD).
   * Burkitt lymphoma:

     * Must have received at least 2 prior lines of therapy
     * Must be ineligible or refuse therapies with demonstrated clinical benefit
   * Follicular lymphoma:

     * Must have received 3 prior lines of therapy, and must have received rituximab and chemotherapy
4. Patients with solid tumors have measurable disease based on RECIST 1.1. In hematological malignancies LYRIC/Lugano will be used.
5. In defined cohorts, patients must have confirmed positive expression of CD161. Patients must have an available archival biopsy sample or agree to have a fresh biopsy obtained to confirm positivity and must agree to a mandatory newly obtained on-treatment biopsy.

Phase 1B:

Must meet all of eligibility criteria in Phase 1, AND the following:

1. Must have histologically or cytologically-documented, unresectable, locally-advanced or metastatic MSS CRC with documented IHC for MMR and/or DNA for MSI consistent with MSS CRC.
2. Eligible for treatment with fruquintinib according to the FDA-approved USPI
3. Must have received no more than 3 lines of systemic therapy for metastatic or unresectable disease, consisting of prior treatment with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if RAS wild-type and medically appropriate, an anti-EGFR therapy. Neoadjuvant or adjuvant systemic therapy is not counted as a prior line, and standard of care agents need not be repeated in the metastatic setting if not clinically indicated in the opinion of the investigator
4. Body weight ≥40kg

Phase 2A:

Inclusion criteria for these patients will remain similar to those used during Phase 1.

Key Exclusion Criteria:

Phase 1:

1. Any prior Grade 4 immune-mediated adverse event (imAE) or Grade 3 imAE requiring steroid treatment (>10 mg/day prednisone or equivalent dose for more than 12 weeks) while receiving immunotherapy that has been documented within the 12 months prior to enrollment.
2. Unresolved toxicity higher than Grade 1 CTCAE v 5 (or higher) attributed to any prior therapy/procedure at screening, except for alopecia.
3. Prior history of serious hypersensitivity reaction to treatment with a monoclonal antibody
4. Patients who are currently pregnant or breastfeeding
5. Use of other investigational drugs (drugs not marketed for any indication) within 14 days or at least 5 half-lives (whichever is shorter) before investigational enrollment (Day 1, Cycle 1 dosing)
6. Patient with history of malignancy (other than the one for which he/she participates in the study or than basal cell carcinoma definitively resected, or other in situ cancers) - unless the patient has undergone curative therapy with no evidence of that disease for 3 years
7. Patients currently receiving cancer therapy (ie, chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery, and/or tumor embolization) or expected to require any other form of antineoplastic therapy while on study.
8. Patients with active, known or suspected autoimmune disease requiring systemic treatment (corticosteroids or other active immunosuppressive medications) within the past 6 months - with the exclusion of vitiligo, resolved asthma/atopia or alopecia areata; hypothyroidism stable on hormone replacement.
9. Known CNS metastases (unless clinically stable for at least 4weeks prior to enrollment and off steroids for at least 7 days- exceptions above for physiologic replacement doses of hydrocortisone)
10. Myocardial infarction, symptomatic congestive heart failure (NYHA> Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of screening
11. Patient has history of or current HIV, Hepatitis B or C infection, even if not active and/or controlled

Phase 1B:

Must not have met any exclusion criteria for Phase 1, and must not have any of the following:

1. Serum electrolytes, potassium, calcium, or magnesium levels outside of the normal laboratory reference range and clinically significant in the investigator's judgment
2. Serum creatinine >1.5 × ULN or creatinine clearance <60 L/min.
3. Urine dipstick protein ≥2+ or 24-hour urine protein ≥1.0 g/24-h
4. Uncontrolled hypertension, defined as: systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg despite optimal medical management
5. History of arterial thromboembolic events within the past 3 months that are not adequately controlled in the opinion of the investigator
6. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction or coronary artery bypass surgery, symptomatic congestive heart failure (New York Heart Association [NYHA] Classification > Class II), severe or unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of screening
7. Patient has history of or current human immunodeficiency virus (HIV), or hepatitis B infection, even if not active and/or controlled. Prior hepatitis C virus (HCV) infection treated with a full course of curative intent antivirals with an undetectable viral load (below the lower limit of detection) are eligible
8. Use of strong inducers or inhibitors of CYP3A4 within 2 weeks prior to the first dose of study drug and while on study
9. Planned major surgery within 2 weeks prior to study start or during the study

Phase 2A:

Exclusion criteria are expected to remain the same as Phase 1 unless there is a need to further refine expansion cohort populations for Phase 2a. Patients must have a CD161 positive tumor demonstrated by the IHC CLIA assay for each analyte.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation - number of participants with dose limiting toxicities (DLTs) from IMT-009 monotherapy | 21 days (Cycle 1 Day 1- Cycle 1 Day 21)
Dose Escalation- Number of participants with adverse events following administration of IMT-009 | From informed consent (Cycle 0 Day -28) to 90 days after the last dose of IMT-009. Each cycle is 21 days
Phase 1b Cohort(s) number of participants with dose limiting toxicities (DLTs) from IMT-009 in combination with fruiquintinib | 28 days (Cycle 1 Day 1- Cycle 1 Day 28)
Phase 1b Cohort(s) - Number of participants with adverse events following administration of IMT-009 in combination with fruiquintinib | From informed consent (Cycle 0 Day -28) through 90 days after last dose of IMT-009. Each cycle is 28 days
Phase 2a Cohort(s) Overall Response Rate (ORR) based on RECIST 1.1 or Lugano criteria (lymphomas only) to assess anti-tumor activity of IMT-009 in each cohort | Every 6 weeks from Cycle 1 Day 1, until disease progression or death or start of a new anti-cancer therapy, up to 2 years. Each cycle is 21 days.

SECONDARY OUTCOMES:
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Area under the plasma concentration-time curve (AUC) of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Maximum plasma concentration (Cmax) of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Minimum plasma concentration (Cmin) of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Volume of distribution (Vd) of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Apparent volume of distribution at steady state determined after intravenous administration (Vss) of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years.Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Terminal half-life (t1/2) of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Time to maximum plasma concentration (Tmax) of IMT-009 when given as monotherapy or in combination | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Pharmacokinetic Analysis: Clearance of IMT-009 when given as monotherapy or in combination. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
  Clearance is the volume of plasma cleared of IMT-009 by the body per unit time.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Number of participants who develop detectable anti-drug antibodies. | Cycle 1 Day 1 to 90 days after treatment discontinuation, up to 2 years.Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE and Phase 1b Cohort(s) - Receptor Occupancy (RO) to determine the target engagement of IMT-009. | Cycle 1 Day 1 to treatment discontinuation, up to 2 years. Dose Escalation and PDE cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE and Phase 1b Cohort(s) - Overall Response Rate (ORR) based on RECIST 1.1 or Lugano criteria (lymphomas only) to assess anti-tumor activity of IMT-009. | Every 6 weeks from Cycle 1 Day 1, until disease progression or death or start of a new anti-cancer therapy, up to 2 years. Dose Escalation and PDE cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Clinical benefit rate (CBR) based on RECIST 1.1 or Lugano criteria (lymphomas only) to assess preliminary anti-tumor activity of IMT-009. | Every 6 weeks from Cycle 1 Day 1, until disease progression or death or start of a new anti-cancer therapy, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Duration of Response (DOR) based on RECIST 1.1 or Lugano criteria (lymphomas only) to assess preliminary anti-tumor activity of IMT-009. | Every 6 weeks from Cycle 1 Day 1, until disease progression or death or start of a new anti-cancer therapy, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Progression-free survival (PFS) based on RECIST 1.1 or Lugano criteria (lymphomas only) to assess preliminary anti-tumor activity of IMT-009. | Every 6 weeks from Cycle 1 Day 1, until disease progression or death or start of a new anti-cancer therapy, up to 2 years. Dose Escalation, PDE and Phase 2a cycles are 21 days. Phase 1b cycles are 28 days.
Dose Escalation, PDE, Phase 1b and Phase 2a Cohort(s) - Overall survival (OS) to assess preliminary anti-tumor activity of IMT-009. | Cycle 1 Day to discontinuation of study drug, then every 3 months for up to 2 years.
Phase 2a Cohort(s)- Number of participants with adverse events following administration of IMT-009. | From informed consent (Cycle 0 Day -28) to 30 days after the last dose of IMT-009. Each cycle is 21 days.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Site 9618, Tucson, Arizona
  - Site 5000, Denver, Colorado
  - Site 4100, Orlando, Florida
  - Site 4060, Sarasota, Florida
  - Site 4500, Oklahoma City, Oklahoma
  - Site 9280, Portland, Oregon
  - Site 3000, Nashville, Tennessee
  - Site 9384, Austin, Texas
  - Site 9112, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No